CLINICAL TRIAL: NCT00696735
Title: Randomized Phase III Study Comparison Between Conventional Chemotherapy and High-Dose Therapy Followed by Autologous Purged Stem-Cell Transplantation in Patients With Follicular Lymphoma Stage III,IV First-Line Treatment for Patients Younger Than 60 Years Old With a High Tumor Burden
Brief Title: High-Dose Therapy Treatment in Patients With Follicular Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: GOELAMS 064 Trial, GOELAMS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOELAMS 064
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2006-09

CONDITIONS: Follicular Lymphoma
Keywords: Phase III study patients with follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Drug Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): standard chemotherapy arm, the CHVP (cyclophosphamide, low-dose doxorubicin, teniposide, and prednisone) regimen consisted of cyclophosphamide (600 mg/m2), doxorubicin (25 mg/m2), and teniposide (60 mg/m2), all administered intravenously on day 1, and prednisone (40 mg/m2), administered orally on days 1 to 5.4,12 Treatment consisted of a 6-course induction phase administered monthly, followed, for responders and patients presenting a stable disease, by a maintenance phase that consisted of 1 cycle every 2 months for 1 year. Concomitant subcutaneous interferon alfa-2b was administered at 5 x 106 3 times a week for 18 months.
  Interventions: Procedure: chemotherapy
- 2 (Experimental): VCAP (cyclophosphamide, high-dose doxorubicin, prednisone, and vincristine) regimen as a first-line therapy combining vindesine (3 mg/m2) on day 1, cyclophosphamide (1500 mg/m2) on day 2, doxorubicin (80 mg/m2) on day 2, and prednisolone (50 mg/m2) on days 1 to 5, every 3 weeks.19,31,32 Patients in CR, VGPR, or PR after the second or third VCAP cycle continued on to stem-cell harvesting and received, before transplantation, one course of IMVP16 (ifosfamide, methotrexate, and VP-16), which combined ifosfamide (1.5 g/m2) and VP16 (100 mg/m2) on days 1 through 3, and methotrexate (30 mg/m2) on days 1 and 10. Patients with less than PR after the VCAP cycles received, as salvage therapy, 2 to 3 courses of DHAP (dexamethasone, high-dose cytarabine, and cisplatin) combining cisplatine (100 mg/m2) on day 1, cytarabine (4 g/m2) on day 2, and dexamethasone (40 mg/m2) on days 1 through 4. If at least a PR was obtained after DHAP, stem cells were harvested or patients were considered as failures
  Interventions: Procedure: high dose therapy and autologous stem cell transplantation

INTERVENTIONS:
Procedure: chemotherapy — injection cyclophosphamide doxorubicin (25 mg/m2), and teniposide (60 mg/m2)(600 mg/m2)on day 1 and prednisone (40 mg/m2), administered orally on days 1 to 5.4,12 Treatment consisted of a 6-course induction phase administered monthly, followed, for responders and patients presenting a stable disease, by a maintenance phase that consisted of 1 cycle every 2 months for 1 year. Concomitant subcutaneous interferon alfa-2b was administered at 5 x 106 3 times a week for 18 months.
  Arms: 1
Procedure: high dose therapy and autologous stem cell transplantation — VCAP regimen 3 cycles , less than PR: 2-3 DHAP, stem cell collection, in vitro purging autologous stem cell transplantation with TBI and cyclophosphamide
  Arms: 2

SUMMARY:
Follicular lymphomas are a subgroup of B-cell non-Hodgkin lymphomas, accounting for 15% to 30% of newly diagnosed lymphomas.1-3 Median survival varies from 5 to 10 years depending on the prognostic factors at diagnosis and response to first-line therapy.4-6 Whatever the treatment, no plateau appears on survival curves, and virtually all patients relapse; follicular lymphomas are ultimately progressive, and fatal.2,3,5 No reference first-line treatment is clearly defined. One of the most active therapies is still doxorubicin-based chemotherapy with or without interferon.7-9 New therapeutic approaches including purine analogs and anti-CD20 monoclonal antibody are promising and are progressively included in the management of these lymphomas.2,3,10-13 The role of high-dose therapy (HDT) as a salvage treatment for patients with relapsing follicular lymphoma is demonstrated by some authors; several reports have shown the superiority of HDT followed by autologous stem-cell transplantation, purged or unpurged, compared with conventional chemotherapy in terms of no relapse and overall survival.14-18 Only a few reports have been published showing HDT results as a first-line treatment for poor-risk patients with follicular lymphoma, and the results remain controversial.19-26 These data prompted the French Groupe Ouest-Est des Leucémies et Autres Maladies du Sang (GOELAMS) to conduct a prospective randomized trial using patients with newly diagnosed follicular lymphoma with a high tumor burden. A combined doxorubicin-based chemotherapy associated with interferon was compared to front-line HDT followed by purged autologous stem-cell transplantation.

DETAILED DESCRIPTION:
Age 8-60 years old follicular lymphoma Not previously treated Stage II bulky, III or IV An Arbor classification high tumor burden

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* Follicular Lymphoma B, C or D (Working Formulation)
* No previous treatment
* Seronegativity HIV
* ECOG performance status less than or 2
* eligible for autologous stem-cell transplantation
* Stage II , III or IV Ann Arbor Classification
* criterias of high tumor burden
* Patient's written informed consent

Exclusion Criteria:

* Age less than 18 years old or more than 60 years old
* Other type of lymphoma
* Stage less than 3 or III-IV (faible masse)
* Seropositivity HIV
* Patients with a history of another malignancy except basal cell skin cancer or in situ uterus cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 1994-06; Primary Completion 2003-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
event free survival | from diagnosis to first event

SECONDARY OUTCOMES:
safety | from diagnosis to death

CONTACTS AND LOCATIONS:
Overall Officials: Philippe COLOMBAT, MD PHD, Principal Investigator — French Innovative Leukemia Organisation
Locations (2):
- France (2):
  - Emmanuel GYAN, Tours
  - Philippe COLOMBAT, Tours

REFERENCES:
- [Derived] Gyan E, Foussard C, Bertrand P, Michenet P, Le Gouill S, Berthou C, Maisonneuve H, Delwail V, Gressin R, Quittet P, Vilque JP, Desablens B, Jaubert J, Ramee JF, Arakelyan N, Thyss A, Molucon-Chabrot C, Delepine R, Milpied N, Colombat P, Deconinck E; Groupe Ouest-Est des Leucemies et des Autres Maladies du Sang (GOELAMS). High-dose therapy followed by autologous purged stem cell transplantation and doxorubicin-based chemotherapy in patients with advanced follicular lymphoma: a randomized multicenter study by the GOELAMS with final results after a median follow-up of 9 years. Blood. 2009 Jan 29;113(5):995-1001. doi: 10.1182/blood-2008-05-160200. Epub 2008 Oct 27. PMID 18955565